CLINICAL TRIAL: NCT00744770
Title: A Phase I, Open-label, Single-sequence Drug-drug Interaction Trial in Subjects on Stable Methadone Maintenance Therapy, to Investigate the Potential Interaction Between TMC278 25 mg q.d. and Methadone, at Steady-state.
Brief Title: TMC278-TiDP6-C121: Drug-drug Interaction Trial to Investigate the Potential Interaction Between TMC278 25 mg Daily and Methadone, at Steady State.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002524
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV
Keywords: TMC278-TiDP6-C121; TMC278-C121; open-label; drug-drug interaction; methadone; TMC278
MeSH Terms: interventions — Rilpivirine

INTERVENTIONS:
Drug: TMC278

SUMMARY:
The purpose of this Phase I, open-label, single-sequence drug-drug interaction trial in patients on stable methadone maintenance therapy is to investigate the potential interaction between TMC278 25 mg daily and methadone, at steady-state.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single-sequence drug-drug interaction trial in patients on stable methadone maintenance therapy, to investigate the potential interaction between TMC278 25 mg daily and methadone, at steady-state. TMC278 is under development for the treatment of HIV-1 infected patients. The trial population will consist of 16 HIV-negative patients on stable methadone maintenance therapy. Patients will receive TMC278 25 mg daily for 11 days, added to their current methadone therapy. The current methadone dosage for each patient is not to be changed from screening until Day 11 inclusive. Methadone dose will be individualized for each patient and should be between 60 and 150 mg daily. Full 24 hour pharmacokinetic profiles of R- and S-methadone will be determined on Day -1 (methadone alone) and on Day 11 (methadone + TMC278). A full 24 hour pharmacokinetic profile of TMC278 will be determined on Day 11 (methadone + TMC278). Pharmacodynamic assessments of the symptoms of methadone withdrawal (Short Opiate Withdrawal Scale (SOWS), Desires for Drugs Questionnaire (DDQ), pupillometry) will be performed on Day -7 and daily from Day -3 until Day 11, within 2 hours before the intake of methadone. Safety and tolerability will be evaluated continuously throughout the trial. Patients will receive TMC278 added to their current methadone therapy in the following way: methadone individualized maintenance therapy, 60 to 150 mg daily from Day -14 to 11 and TMC278 25 mg tablet by mouth daily from Day 1 to 11. TMC278 and methadone will both be taken within 10 minutes after completion of a breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 18.0 to 30.0 kg/m2, extremes included
* Receiving once daily oral methadone maintenance therapy at a stable individualized dose of 60 to 150 mg
* The patient agrees not to change the current methadone dose from screening until Day 11 included and to have a daily observed and documented methadone intake from Day -14 until Day 12, and a daily observed and documented TMC278 intake from Day 1 until Day 11
* Able to comply with protocol requirements
* The patient has obtained approval from his/her addiction physician for participation in this trial. Furthermore, the addiction physician agrees to provide medical care for the patient after discharge from the testing facility
* General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial
* Otherwise healthy on the basis of a physical examination, medical history (except drug abuse), ECG, vital signs and the results of blood biochemistry and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* A positive test for HIV-1, HIV-2, hepatitis A virus or hepatitis B virus
* female of child bearing potential
* evidence of current use of illicit drugs or opioids (with the exception of methadone) or abuse of alcohol
* impaired liver function as defined in the protocol
* other currently active or underlying disorders, including gastrointestinal, cardiovascular, neurologic, psychiatric (other than drug dependency), metabolic, adrenal, renal, hepatic, respiratory, inflammatory, or infectious disease
* presence of risk factors for QTc prolongation
* any history of significant skin disease or allergies, including allergy or hypersensitivity to the excipients of the investigational medication TMC278 or to methadone
* Previous experience of clinically significant hypersensitivity to methadone hydrochloride
* Use of disallowed concomitant therapy during the 14 days prior to the first dose of TMC278
* recent donation of blood or plasma or participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of steady-state TMC278 25 mg q.d. on the steady-state pharmacokinetics of R- and S-methadone after 11 days of TMC278 intake.

SECONDARY OUTCOMES:
To evaluate after 11 days of TMC278 intake: the potential effect of TMC278 on the pharmacodynamic effects of methadone therapy; the steady-state pharmacokinetics of TMC278 25 mg daily; the short-term safety and tolerability of coadministration.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Crauwels HM, van Heeswijk RP, Vandevoorde A, Buelens A, Stevens M, Hoetelmans RM. The effect of rilpivirine on the pharmacokinetics of methadone in HIV-negative volunteers. J Clin Pharmacol. 2014 Feb;54(2):133-40. doi: 10.1002/jcph.222. Epub 2013 Nov 23. PMID 24203510